CLINICAL TRIAL: NCT02351466
Title: Type 1 Diabetes and the Brain in Children: Metabolic Interventions. Protocol #1: Longitudinal Assessment
Brief Title: Type 1 Diabetes and the Brain in Children
Status: Completed | Type: Observational
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Stanford University (Other); Washington University School of Medicine (Other); Yale University (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Nelly Mauras, MD, Nemours Children's Clinic
Other Study IDs: 588973
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Brain Growth and Development; Cognition; Children; Continuous Glucose Monitoring; MRI; Functional MRI
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Children with Type 1 Diabetes: Subjects with T1 diabetes will undergo a physical exam and blood test as well as structural and functional brain MRI, neurocognitive testing and wear a continuous glucose monitor every 3 months for 24 months.
  Interventions: Other: Observational
- Healthy Controls: Subjects will undergo a physical exam and blood test as well as structural and functional brain MRI at baseline and after 24 months.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
The investigators have previously studied a group of young children with T1D using brain MRI, age-appropriate neurocognitive testing and continuous glucose monitoring, followed for 18 months. The investigators observed significant differences in gray matter volumes and white matter microstructure in the children with diabetes as compared to controls. These differences appeared to increase over time, with slower rates of brain growth in the T1D group (Mazelli, et al, Diabetes 2014; Barnea-Goraly, et al, Diabetes Care 2014; Mauras, et al, Diabetes 2015). In this new protocol the investigators will include the same children with T1D and healthy controls previously studied and recruit new similar subjects to replace those lost by attrition. The investigators will be using structural and functional brain MRI, neurocognitive testing and measures of glycemic control, to determine if changes in the brain persist or worsen over longitudinal follow up, and whether these changes are associated with measures of glycemic control and neurocognitive metrics as these children grow and progress through puberty.

DETAILED DESCRIPTION:
Study participation will last about 2 to 2 1/12 years and will include a brain MRI without sedation, as well as a functional MRI and neurocognitive testing. The children with T1D will wear a continuous glucose monitor (CGM), will follow up every 3 months and will be asked to wear the CGM each time. The structural and functional MRI and neurocognitive testing will be repeated 2 yrs from baseline.

The healthy controls will also undergo MRI and cognitive testing as well as have a blood sample at baseline and after 2 years.

Parents of newly recruited subjects will also have abbreviated IQ testing.

ELIGIBILITY:
Inclusion Criteria for T1 Diabetes Group:

* Diabetes diagnosed after age 6 months
* Gestational age >34 weeks, birth weight >2kg

Inclusion Criteria for Healthy Control Group:

* Normal HbA1C and fasting blood glucose
* Negative diabetes auto-antibodies (those that are siblings of T1D patients)
* Gestational age >34 weeks, birth weight >2kg

Exclusion Criteria for Both Groups:

* History of mental retardation, language or learning disability
* Known genetic or medical problem that could impair brain development
* Abnormality of the brain/nervous system, visual or hearing problem
* History of seizures not associated with fever
* Previous inpatient psychiatric treatment
* Unable to have a MRI of the head due to metal appliances

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with Type 1 Diabetes or Healthy non-diabetic controls
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2015-03; Primary Completion 2018-11 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Changes in total and regional gray and white matter volumes and white matter microstructure. | 2 years
  Structural MRIs of children with T1 diabetes will be compared to age- and sex-matched, non-diabetic healthy controls. We will investigate whether these changes are associated with measures of glycemic control and neurocognitive metrics as these children grow and progress through puberty. The present cohorts (T1D and controls) of young children will be followed for 2 more years with similar studies repeated 2 years apart. Overall glycemic profiles will continue to be obtained every 3 months longitudinally between scans with CGM and HbA1c for children with Type 1 Diabetes.

SECONDARY OUTCOMES:
Measures of activation of frontal-parietal networks and functional connectivity of resting state networks using blood oxygen level dependent (BOLD)-functional MRI. | 2 years
Changes in Neurocognitive metrics including IQ as well as executive and visual-spatial memory. | 2 years
  We will perform neurocognitive metrics reflecting frontal, parietal-occipital and hippocampal function. Children with T1D will be followed longitudinally and compared with controls to determine whether these differences are associated with measures of glycemic control.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Mauras, MD, Principal Investigator — Nemours Children's Clinic; Allan L Reiss, MD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Nemours Childrens Clinic, Jacksonville, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Washington University, St Louis, Missouri

REFERENCES:
- [Background] Mauras N, Mazaika P, Buckingham B, Weinzimer S, White NH, Tsalikian E, Hershey T, Cato A, Cheng P, Kollman C, Beck RW, Ruedy K, Aye T, Fox L, Arbelaez AM, Wilson D, Tansey M, Tamborlane W, Peng D, Marzelli M, Winer KK, Reiss AL; Diabetes Research in Children Network (DirecNet). Longitudinal assessment of neuroanatomical and cognitive differences in young children with type 1 diabetes: association with hyperglycemia. Diabetes. 2015 May;64(5):1770-9. doi: 10.2337/db14-1445. Epub 2014 Dec 8. PMID 25488901
- [Background] Cato MA, Mauras N, Ambrosino J, Bondurant A, Conrad AL, Kollman C, Cheng P, Beck RW, Ruedy KJ, Aye T, Reiss AL, White NH, Hershey T; Diabetes Research in Children Network (DirecNet). Cognitive functioning in young children with type 1 diabetes. J Int Neuropsychol Soc. 2014 Feb;20(2):238-47. doi: 10.1017/S1355617713001434. PMID 24512675
- [Background] Barnea-Goraly N, Raman M, Mazaika P, Marzelli M, Hershey T, Weinzimer SA, Aye T, Buckingham B, Mauras N, White NH, Fox LA, Tansey M, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Alterations in white matter structure in young children with type 1 diabetes. Diabetes Care. 2014 Feb;37(2):332-40. doi: 10.2337/dc13-1388. Epub 2013 Dec 6. PMID 24319123
- [Background] Marzelli MJ, Mazaika PK, Barnea-Goraly N, Hershey T, Tsalikian E, Tamborlane W, Mauras N, White NH, Buckingham B, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Neuroanatomical correlates of dysglycemia in young children with type 1 diabetes. Diabetes. 2014 Jan;63(1):343-53. doi: 10.2337/db13-0179. Epub 2013 Oct 29. PMID 24170697
- [Background] Barnea-Goraly N, Weinzimer SA, Ruedy KJ, Mauras N, Beck RW, Marzelli MJ, Mazaika PK, Aye T, White NH, Tsalikian E, Fox L, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). High success rates of sedation-free brain MRI scanning in young children using simple subject preparation protocols with and without a commercial mock scanner--the Diabetes Research in Children Network (DirecNet) experience. Pediatr Radiol. 2014 Feb;44(2):181-6. doi: 10.1007/s00247-013-2798-7. Epub 2013 Oct 6. PMID 24096802
- [Background] Tansey M, Beck R, Ruedy K, Tamborlane W, Cheng P, Kollman C, Fox L, Weinzimer S, Mauras N, White NH, Tsalikian E; Diabetes Research in Children Network (DirecNet). Persistently high glucose levels in young children with type 1 diabetes. Pediatr Diabetes. 2016 Mar;17(2):93-100. doi: 10.1111/pedi.12248. Epub 2014 Dec 11. PMID 25496062
- [Derived] Mauras N, Buckingham B, White NH, Tsalikian E, Weinzimer SA, Jo B, Cato A, Fox LA, Aye T, Arbelaez AM, Hershey T, Tansey M, Tamborlane W, Foland-Ross LC, Shen H, Englert K, Mazaika P, Marzelli M, Reiss AL; Diabetes Research in Children Network (DirecNet). Impact of Type 1 Diabetes in the Developing Brain in Children: A Longitudinal Study. Diabetes Care. 2021 Apr;44(4):983-992. doi: 10.2337/dc20-2125. Epub 2021 Feb 10. PMID 33568403